CLINICAL TRIAL: NCT07381972
Title: Optimization of Photodynamic Therapy Through the Association With Sonodynamic Therapy for the Treatment of Nodular Basal Cell Carcinoma
Brief Title: Photodynamic Therapy Associated With Sonodynamic Therapy for the Treatment of Nodular Basal Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Gabriela Salvio, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7.810.244; U1111-1330-4954 (Other: UTN (Universal Trial Number))
Record Dates: First submitted 2026-01-13; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Nodular Basal Cell Carcinoma of Skin
Keywords: Photodynamic Therapy; Sonodynamic Therapy; Non-melanoma skin cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photodynamic therapy (PDT) protocol (Active Comparator): In this arm, lesions will be treated with the conventional PDT protocol for this type of lesion.
  Interventions: Combination Product: Control Arm (Conventional Therapy)
- Sono-Photodynamic Therapy (SonoPDT) protocol (Experimental): In this arm, lesions will be treated with a modified treatment protocol called SonoPDT protocol.
  Interventions: Combination Product: Experimental arm

INTERVENTIONS:
Combination Product: Control Arm (Conventional Therapy) — PDT protocol: This intervention consists of two therapeutic sessions performed on the same day. The first session involves the application of MAL (methyl aminolevulinate) cream to the skin tumor, followed by an incubation period of 3 hours. After this time, the lesion is illuminated for 20 minutes at an irradiance of 125 mW/cm² using the LINCE device. Following the illumination procedure, the second session begins with a new application of MAL cream and an additional 1.5 hours of incubation. After this period, illumination is performed using the same light parameters as in the first session. After each MAL application, an occlusive dressing composed of PVC film, aluminum foil, gauze, and adhesive tape is applied to the lesion area to prevent light exposure and degradation of the produced PpIX.
  Arms: Photodynamic therapy (PDT) protocol
Combination Product: Experimental arm — SonoPDT protocol: This intervention consists of two therapeutic sessions performed on the same day. The first session involves the application of MAL (methyl aminolevulinate) cream to the skin tumor, followed by an incubation period of 3 hours. After this time, the lesion is illuminated for 20 minutes at an irradiance of 125 mW/cm² using the LINCE device. Immediately after illumination, the lesion will be irradiated with ultrasound (frequency: 1MHz, mode: pulsed, ultrasound intensity: 1.5 W/cm2, duty cycle: 50%, pulse frequency: 100 Hz) for 5 minutes. Following the sonication procedure, the second session begins with a new application of MAL cream with an incubation period of 1.5 hours. After this time, illumination and sonication are performed using the same excitation source parameters as in the first session.
  Arms: Sono-Photodynamic Therapy (SonoPDT) protocol

SUMMARY:
Evaluation of a therapeutic protocol based on the combination of photodynamic therapy and sonodynamic therapy, referred to as sonophotodynamic therapy. Since this new protocol is applied in a single day, it is called the single-visit Sono-PDT protocol. This protocol will be used for the treatment of nodular basal cell carcinoma lesions.

DETAILED DESCRIPTION:
In the proposed treatment protocol, all the procedures of traditional PDT protocol will be maintained, with the addition of a dose of low-intensity therapeutic ultrasound immediately after the application of red light. Ultrasound, due to its greater ability to penetrate the skin, can help reach deeper tumor cells and thus improve treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, aged 18 years and older.
* Histologically confirmed nodular basal cell carcinoma with lesion diameter ≤1.0 cm.
* Participants with multiple lesions may be included, provided that each lesion meets all inclusion criteria.

Exclusion Criteria:

* Nodular basal cell carcinoma lesions >1.0 cm in diameter.
* Known hypersensitivity or allergy to methyl aminolevulinate (MAL) or any excipients of the study medication.
* Histological subtypes of infiltrative basal cell carcinoma, including micronodular, infiltrative, sclerodermiform (morpheaform), plano-cicatricial, or terebrant subtypes.
* Porphyria or other disorders of porphyrin metabolism.
* Pregnant or breastfeeding women.
* Women of childbearing potential not using an acceptable method of contraception.
* Presence of photosensitive diseases, including lupus erythematosus.
* Any condition that, in the investigator's opinion, would interfere with study participation or safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the complete response rate after one month of treatment. | One month after the treatment was applied to the patient.
  Complete response will be defined as the absence of clinical and/or histopathological signs of the tumor after one month of treatment.

SECONDARY OUTCOMES:
Evaluation of the complete response rate and recurrence-free survival rate after six months of treatment. | Six months after the treatment was applied to the patient.
  Complete response will be defined as the absence of clinical and/or histopathological evidence of the tumor. Recurrence-free survival at 6 months will be determined by the proportion of patients who show no recurrence of the lesion at the treated site or in adjacent areas within 6 months, relative to the total number of patients treated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Amaral Carvalho, Jaú, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayala ETP, Carvalho ISE, Antunes CA, Mahmood A, Requena MB, Alves F, Pires L, Yakovlev V, Bagnato VS, Pratavieira S. Comparative analysis of ALA mediated sonodynamic therapy considering tumor size, light combination and ultrasound delivery in murine cutaneous melanoma. Sci Rep. 2025 Aug 22;15(1):30859. doi: 10.1038/s41598-025-16366-x. PMID 40846765
- [Background] Salvio AG, Veneziano DB, Moriyama LT, Inada NM, Grecco C, Kurachi C, Bagnato VS. A new photodynamic therapy protocol for nodular basal cell carcinoma treatment: Effectiveness and long-term follow-up. Photodiagnosis Photodyn Ther. 2022 Mar;37:102668. doi: 10.1016/j.pdpdt.2021.102668. Epub 2021 Dec 1. PMID 34863948